CLINICAL TRIAL: NCT06091566
Title: Safety and Performance of UCon Bar Electrode for the Treatment of Overactive Bladder (OAB) and Bowel Dysfunction (BD) - An Early Feasibility Study
Brief Title: Safety and Performance of UCon Bar Electrode for the Treatment of Overactive Bladder (OAB) and Bowel Dysfunction (BD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InnoCon Medical (Industry)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK_FEAS_02
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Urge; Fecal Incontinence; Fecal Incontinence With Fecal Urgency; Nocturia; Urinary Frequency More Than Once at Night; Bowel Disorders Functional; Incontinence, Nighttime Urinary
Keywords: Urinary Incontinence; Fecal Incontinence; Urge incontinence; Neurostimulation; Dorsal Genital Nerve
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Fecal Incontinence; Nocturia; Nocturnal Enuresis

STUDY DESIGN:
Intervention Model Description: Single-group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrical stimulation (Experimental): Electrical stimulation to the dorsal genital nerve.
  Interventions: Device: UCon-Bar

INTERVENTIONS:
Device: UCon-Bar — The participant self-administer electrical stimulation to the dorsal genital nerve (DGN) for either 4 weeks or 12 weeks using UCon with the Bar electrode
  Other Names: Electrical stimulation to the dorsal genital nerve (DGN stimulation)

SUMMARY:
UCon is a medical device for treatment of the symptoms of overactive bladder (OAB) and bowel dysfunction (BD). It electrically stimulates the DGN through the skin to obtain modulated behaviour of the bladder/bowel musculature e.g., suppress undesired bladder/bowel activity to relieve the symptoms of the patient.

This clinical investigation is designed as a single-arm, prospective, multi-centre, and early feasibility study.

DETAILED DESCRIPTION:
The overall purpose of the current clinical investigation is to evaluate the medical device with a UCon-Bar Electrode with respect to its initial safety and device performance in a cohort of 40 female patients with OAB/BD over a period of 12 weeks.

The investigation consists of two periods: a screening period and an intervention period.

During the screening period, the participants will be using UCon with a Patch Electrode and complete a 4 week stimulation period at home. The screening period will determine if participants fulfil the criteria to participate in the intervention period.

During the intervention period, the UCon Bar Electrode will be inserted in the clitoral hood. After a recovery period (4-8 weeks), the participants will be using UCon with the Bar Electrode and complete wither a 4 week or a 12 week stimulation period at home.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is female
2. Participant is ≥ 18 years of age.
3. Participant is diagnosed with OAB or BD.

   OAB: Urinary urgency usually with one or more of the following:

   i. Urinary urgency incontinence (≥1 per/week). ii. Urinary frequency (≥8 voiding/day without polyuria). iii. Nocturia (≥2 voiding/night without nocturnal polyuria).

   BD: One or more of the following:

   i. Faecal urgency (≥3 urgencies pr. week) together with registration of urgency in St. Mark´s and a St. Mark´s score ≥9.

   ii. Faecal incontinence (urge/passive) (≥1 per/week).
4. Participant is able to communicate, provide feedback, understand and follow instructions during the course of the investigation, including using the device at home.

Exclusion Criteria:

1. Participant is medically unstable (acute illness or complication of a chronic condition, apart from the OAB or BD, that might affect the participants´ participation in the investigation).
2. Participant has an active infection in the genital area.
3. Participant has an implanted pacemaker, implantable drug pump or other active medical devices (any medical device that uses electrical energy or other sources of power to make it function).
4. Participant is pregnant, nursing or planning a pregnancy (to be confirmed with a negative pregnancy test). Women of childbearing potential must maintain effective contraception during the clinical investigation.
5. Participant is enrolled or planning to enrol in another conflicting clinical investigation or was enrolled in an investigational drug trial or medical device investigation within four weeks of enrolment.
6. Participant has neuropathy to a degree that is presumed to diminish the effect of the electrical stimulation.
7. Participant has a history of cancer in the pelvic region, are currently receiving cancer treatment, or has received radiation therapy in the pelvic region.
8. Participant has addictive behaviour defined as the abuse of alcohol, cannabis, opioids, or other intoxicating drugs.
9. Participant does not speak or understand Danish.

   * The following contraception is considered effective: Intrauterine device, hormonal contraceptives such as birth control pills, implants, contraceptive patch, vaginal ring, and contraceptive injection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
PRIMARY SAFETY: ratio of participants with successful insertion of the UCon Bar Electrode. | After 4 weeks and 12 weeks
  1) Number and severity of adverse events during insertion of the UCon Bar Electrode: Excessive pain and excessive bleeding. 2) Number and severity of adverse events after insertion: Infection, pain, and bleeding. 3) Number of participants with successful insertion with no premature removal of the Bar Electrode.
PRIMARY PERFORMANCE: ratio of treatment change [performance] of OAB/BD symptoms | Change from baseline at 4 weeks and/or 12 weeks
  Ratio of participants with at least 50% reduction of their OAB/BD symptoms from baseline as assessed by subjective reporting in an electronic bladder or bowel diary.

SECONDARY OUTCOMES:
SECONDARY SAFETY: Characterization, including frequency and severity of adverse events related to the risks and anticipated adverse device effects associated with the use of UCon-Bar Electrode. | After 4 weeks and 12 weeks
  1) Characterization of adverse events and adverse device effects associated with the use of UCon-Bar during the investigational period.2) Number of participants experiencing adverse events and adverse device effects associated with the use of UCon-Bar during the investigational period.3) Number and severity of adverse events and adverse device effects associated with the use of UCon-Bar during the investigational period.
SECONDARY PERFORMANCE: ratio of treatment change [performance] of OAB/BD symptoms | Change from baseline at 4 weeks and/or 12 weeks
  Ratio of participants with at least 33% reduction of their OAB/BD symptoms from baseline as assessed by subjective reporting in an electronic bladder or bowel diary.
SECONDARY PERFORMANCE: assess whether participants using UCon Bar Electrode experience a change in their quality of life | Change from baseline at 4 weeks and/or 12 weeks
  Ratio of subjects with a change in their self-reported quality of life measures as assessed by specific QoL questionnaires related to OAB (ICIQ-OAB, an overall score with greater values indicates increased symptom severity) or BD (St. Marks incontinence score and Rockwood Fecal Incontinence Quality of Life Scale, an overall score with greater values indicates a worse symptom outcome.)
SECONDARY PERFORMANCE: assess whether participants using UCon Bar Electrode experience an impression of treatment improvement | After 4 week screening period, 4 weeks, and 12 weeks
  Ratio of participants with a self-reported improvement in their impression of treatment as assessed by the 7-point Patient Global Impression of Improvement (PGI-I) scale. An improvement is defined as choosing one of the following: very much, better, much better, or a little better.
SECONDARY PERFORMANCE: ratio of participant that accept UCon and DGN stimulation [Device and treatment acceptability of UCon] | After 4 week screening period, 4 weeks, and 12 weeks
  Ratio of participants that accept UCon and DGN stimulation as assessed by a satisfaction survey recorded after each stimulation periods (with UCon Patch Electrode and UCon Bar Electrode) .
Secondary PERFORMANCE: ratio of treatment change [performance] of OAB/BD symptoms during the screening period can be reproduced in the intervention period. | Change from screening period at 4 weeks and/or 12 weeks
  Ratio of participants with at least 50% reduction in symptoms using the UCon-Patch Electrode, that can be reproduced in 80% of the participants using the UCon Bar Electrode.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Christensen, MD, Principal Investigator — Palle Juul Jensens Boulevard 99 DK-8200 Aarhus N
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No